CLINICAL TRIAL: NCT06251427
Title: Assessing the Effectiveness of a Multiple-micronutrient Fortified Maize Pap on the Nutrient Status of Nigerian School-aged Children: Randomized Controlled Trial
Brief Title: Assessing the Effectiveness of a Multiple-micronutrient Fortified Maize Pap on the Nutrient Status of Nigerian School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Collaborators: University of Ibadan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Aladdin
Record Dates: First submitted 2024-01-17; First posted 2024-02-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Iron Deficiencies
Keywords: School-aged children; Nigeria; Multiple-micronutrient fortification; School feeding program
MeSH Terms: conditions — Iron Deficiencies | interventions — Milk

STUDY DESIGN:
Intervention Model Description: Three armed double blinded intervention.
  1. Low dose of multiple micronutrient fortification
  2. Moderate dose of multiple micronutrient fortification
  3. High dose of multiple micronutrient fortification
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose multiple micronutrient fortification (Placebo Comparator): Maize, milk plus low multiple micronutrient fortification
  Interventions: Dietary Supplement: Multiple micronutrient fortified maize with milk
- Moderate dose multiple micronutrient fortification (Active Comparator): Maize, milk plus moderate multiple micronutrient fortification
  Interventions: Dietary Supplement: Multiple micronutrient fortified maize with milk
- High dose multiple micronutrient fortification (Active Comparator): Maize, milk plus high multiple micronutrient fortification (double the moderate level)
  Interventions: Dietary Supplement: Multiple micronutrient fortified maize with milk

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient fortified maize with milk — The study product is a multiple micronutrient fortified maize pap with milk

SUMMARY:
A new product was developed by FrieslandCampina for Sub-Saharan Africa as affordable nutrition to nourish Nigerian families of low to middle-socioeconomic class (SEC). It can potentially be used to enhance the ongoing school feeding programs, which are aimed at reducing malnutrition, including micronutrient deficiencies. The main component of the product is maize, which is a traditional staple in Nigeria. The product also contains milk (being a good source of high quality protein) fortified with various micronutrients including iron, iodine, zinc, vitamin A and vitamin B12 at levels contributing to approximately 1/3 of daily recommended intakes per serving of product. Intake of this product may therefore contribute to improvement of micronutrient status among Nigerian schoolchildren suffering from such nutrient deficiencies. Micronutrients are important for various processes in the body, which in turn may influence other outcomes as cognitive performance, reduce illness and improve growth.

DETAILED DESCRIPTION:
The study is a double-blinded three-arm intervention trial. The individual children will be randomised into the three different arms of the study, with varying doses of micronutrients (1) low, (2) medium and (3) high.

The 50g of study product will be given to school children every school day (5/7 days of the week) for 5 intervention months.

Study product: A fermented maize pap, with soy, dairy and multiple micronutrient fortification. Active components: Multiple micronutrient fortification, including ferrous fumarate. Amount of micronutrients differ based on the arm of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Nigerian children in primary schools, aged 5-8 years
2. Willing and able to consume the supplied servings of the study product/s or provided control pap
3. Having written and oral informed consent from the parent/legal guardian and the participants gave oral and/or written assent.

Exclusion Criteria:

1. Children suffering from severe malnutrition and/or micronutrient deficiencies defined as (such children will be referred to a nearby health centre for appropriate treatment).

   1. Children with Height-for-age (HAZ) and Weight-for-age (WAZ) <- 3 Standard Deviation (SD)
   2. Children showing clinical signs of severe (chronic) anemia i.e. visibly pale, jaundice and lethargic.
2. Children with a history of or who at the time of recruitment suffer from chronic illness, including (but not limited to) renal diseases, thyroid disease, (metabolic) bone disease, genetic and/or congenital disorders e.g. Down syndrome and sickle cell anaemia, hepatic dysfunction, thalassemia or chronic diarrhea (e.g. irritable bowl syndrome). Based on medical history examination.
3. Children with a physical disability or handicap that prevents participation in the study.
4. Children with food allergies or intolerances.
5. Children participating in any other clinical research (or having participated in any such study in the previous half year).
6. Children or a child's family who are intending to withdraw from school or move out of the study region within the study period.
7. Children consuming prescribed 'iron/folic acid, and (multi-)vitamin, and mineral supplements' during the course of the study within the last 2 months prior to the study as a minimum.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 934 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Iron status | 5 months
  There will be a change between the two test groups and the control group in iron status as measured by in hemoglobin (whole blood) g/L .
Serum ferritin | 5 months
  There will be a change between the two test groups and the control group in iron status as measured by serum ferritin (ug/L).

SECONDARY OUTCOMES:
Iron deficiency, iron deficiency anaemia and anemia | 5 months
  There will be a difference in prevalence of iron-deficiency, iron-deficiency anaemia and anaemia, taking modifying factors like soluble transferrin receptor and inflammation markers in plasma into account.
Nutrient status | 5 months
  A difference in nutrient status of selected nutrients (iodine, vitamin A, zinc, vitamin B12, vitamin D)

OTHER OUTCOMES:
Cognitive performance | 5 months
  A difference in cognitive performance score, measured via attention (Digit span backward) and short-term memory (digit-span forward) score (higher scores indicate a better outcome.
Anthropometric scores | 5 months
  Difference in anthropometric status between study arms as measured by height-for-age Z score (HAZ) and weight-for-age (WAZ).
Illness | 5 months
  Difference in morbidity/illness as measured by the reduced frequency of illness over the 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- FrieslandCampina Research and Development, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided